CLINICAL TRIAL: NCT00158483
Title: Anti-Herpetic Treatment Associated With Syndromic Management of Genital Ulcer in Africa: Clinical and Biological Evaluation on HIV-1 and HSV-2 Shedding (ANRS 1212)
Brief Title: Anti-Herpetic Treatment of Genital Ulcer : Effect on HIV & Herpes Shedding (ANRS 1212)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANRS 1212
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Ulcer; Herpes Genitalis
Keywords: Genital herpes; Cofactors of sexual transmission; Syndromic treatment; Genital viral load; Ulcer
MeSH Terms: conditions — Ulcer; Herpes Genitalis | interventions — Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Acyclovir (ACV)

SUMMARY:
Herpes virus type 2 (HSV-2) infection - as a cofactor of human immunodeficiency virus (HIV) transmission - can be targeted by anti-herpetic specific drugs, either as a continuous prophylactic treatment during its asymptomatic shedding phase, or as an episodic treatment during clinically-apparent genital ulcerations. The main objective of this trial will be to demonstrate that acyclovir treatment given during clinical episodes (primary infection or recurrences) can reduce genital shedding of HIV, thereby contributing to a reduction of HIV infectiousness of dually infected individuals (HIV+/HSV+).

DETAILED DESCRIPTION:
Objectives. The proposed project is a randomised placebo-controlled, double-blinded, multicentric therapeutic trial evaluating the association of antiherpetic treatment to the syndromic treatment for the management genital ulcers in Africa, and its impact on the genital shedding of HIV and of Herpes simplex hominis type 2 (HSV-2) virus.

Background. Recent epidemiological studies have shown that infection with HSV-2 is highly prevalent in sub-Saharan Africa, and that HSV-2 seropositivity is a marker of high-risk sexual behaviour. HSV-2 infection is increasingly being recognised as one of the commonest causes of genital ulceration in many African countries. HSV-2 infection may act as a major cofactor for HIV transmission, a fact that has long been underestimated. First, genital ulcers (caused by HSV-2) are by themselves cofactors of HIV transmission, either by increasing infectiousness of dually infected individuals (HSV+/HIV+), or by increasing susceptibility of the seronegative partner. Second, HSV-2 infection may transactivate in vivo the genital replication of HIV, thereby increasing the infectiousness of dually infected individuals.

Rationale and main objective. HSV-2 infection - as a cofactor of HIV transmission - can be targeted by anti-herpetic specific drugs, either as a continuous prophylactic treatment during its asymptomatic shedding phase, or as an episodic treatment during clinically-apparent genital ulcerations. The main objective of this trial will be to demonstrate that acyclovir treatment given during clinical episodes (primary infection or recurrences) can reduce genital shedding of free- or cell-associated HIV, thereby contributing to a reduction of HIV infectiousness of dually infected individuals (HIV+/HSV+). Given the present state of knowledge and hypotheses formulated around the possible role of HSV on the HIV epidemic in Africa, the proposed research will contribute to confirm or invalidate the existence of mutual reinforcement of HSV and HIV replication. This will represent a study of biological plausibility for such an in vivo interaction. In addition the chosen intervention strategy has practical and operational implications in that it will allow the evaluation of a novel approach to syndromic management of genital ulcers in Africa that could later lead to revisions of management guidelines.

Methods. Approximately 600 women presenting with genital ulcers will be enrolled over two years and in two sites: Bangui (Central African Republic) and Accra (Ghana). The syndromic management of patients will include antibiotics to cover the presumptive bacterial causes of genital ulcerations in these settings (chancroid and syphilis), according to national and international guidelines (CDC, UK national guidelines, WHO). In addition, women will be randomised to receive either antiherpetic treatment (acyclovir 400 mg 3 times daily for 5 days, according to UK national guidelines - a shorter regimen than US guidelines) or placebo (similar frequency and duration). Clinical examination and cervicovaginal samplings will be carried out at D0 and at each follow up visit at D2, D4, D7, D14 & D28. These samples will be tested for: etiological diagnosis of ulcers by multiplex PCR; measurement of HIV genital viral loads (measuring free RNA and cell-associated proviral DNA) and HSV-2 DNA genital load; and diagnosis of other common STDs (at D0). Blood samples will be collected at D0, D2 and D28 for HIV, syphilis and HSV-2 serological assays, and for HIV plasma loads as well as CD4 measurements.

The main outcome will be the determination of the impact of anti-herpetic treatment on HIV genital load (and as a corollary, on HSV2 genital load). It will also be possible to measure the impact of antibiotic treatment on HIV viral load. The study will allow to evaluate the validity of novel syndromic treatment approaches for genital ulcer disease, and a long term outcome may be the necessary revision of syndromic management guidelines for GUD to potentially include anti-herpetic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed ulcer
* Resident of city or planning to stay for 1 month
* Be a women

Exclusion Criteria:

* Pregnant women
* Menstruating women
* Positive protein urine test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2003-05; Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Difference of HIV-1 RNA and DNA shedding assessed by performing cervicovaginal lavage (CVL) HIV viral load, among groups
Difference of HSV-2 DNA shedding among groups

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Belec, Study Chair — HEGP, Paris; Gérard Grésenguet, Principal Investigator — Faculté de Médecine Université de Bangui; Philippe Mayaud, Study Chair — London School of Hygiene and Tropical Medecine
Locations (3):
- Centre MST/SIDA, Bangui, Central African Republic
- Ghana (2):
  - WAPTCAS, Accra
  - Kumasi Hospital, Service d'infectiologie, Kumasi

REFERENCES:
- [Background] Legoff J, Bouhlal H, Gresenguet G, Weiss H, Khonde N, Hocini H, Desire N, Si-Mohamed A, de Dieu Longo J, Chemin C, Frost E, Pepin J, Malkin JE, Mayaud P, Belec L. Real-time PCR quantification of genital shedding of herpes simplex virus (HSV) and human immunodeficiency virus (HIV) in women coinfected with HSV and HIV. J Clin Microbiol. 2006 Feb;44(2):423-32. doi: 10.1128/JCM.44.2.423-432.2006. PMID 16455895
- [Background] LeGoff J, Mayaud P, Gresenguet G, Weiss HA, Nzambi K, Frost E, Pepin J, Belec L; ANRS 12-12 Study Group. Performance of HerpeSelect and Kalon assays in detection of antibodies to herpes simplex virus type 2. J Clin Microbiol. 2008 Jun;46(6):1914-8. doi: 10.1128/JCM.02332-07. Epub 2008 Apr 2. PMID 18385443
- [Derived] Mayaud P, Legoff J, Weiss HA, Gresenguet G, Nzambi K, Bouhlal H, Frost E, Pepin J, Malkin JE, Hayes RJ, Mabey DC, Belec L; ANRS 1212 Study Group. Impact of acyclovir on genital and plasma HIV-1 RNA, genital herpes simplex virus type 2 DNA, and ulcer healing among HIV-1-infected African women with herpes ulcers: a randomized placebo-controlled trial. J Infect Dis. 2009 Jul 15;200(2):216-26. doi: 10.1086/599991. PMID 19530940